CLINICAL TRIAL: NCT07045701
Title: Efficacy and Safety of FMXIN002 Epinephrine Powder Nasal Spray for the Treatment of Acute Allergic Reactions in Patients at Risk of Anaphylaxis
Brief Title: FMXIN002 in Patients at Risk of Anaphylaxis
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nasus Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP-009-Epinephrine
Record Dates: First submitted 2025-06-08; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Anaphylaxis Food
MeSH Terms: interventions — Epinephrine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMXIN002 4mg + saline IM (Experimental): Epinephrine powder nasal spray together with a placebo IM injection
  Interventions: Combination Product: Epinephrine 4mg nasal powder spray
- Adrenaline 0.5mg IM + placebo nasal spray (Active Comparator): Epinephrine IM injection together with a placebo nasal spray
  Interventions: Combination Product: Adrenalin 0.5mg Injectable Product

INTERVENTIONS:
Combination Product: Epinephrine 4mg nasal powder spray — Epinephrine nasal powder spray in a unidose nasal applicator device. Will be administered together with a placebo saline IM injection
  Other Names: FMXIN002
  Arms: FMXIN002 4mg + saline IM
Combination Product: Adrenalin 0.5mg Injectable Product — Epinephrine 0.5mg for IM injection. Will be administered together with a placebo nasal powder spray.
  Arms: Adrenaline 0.5mg IM + placebo nasal spray

SUMMARY:
Study Objective To evaluate the efficacy of FMXIN002, a powder-based intranasal epinephrine spray, for treating anaphylaxis.

Study Design

• Hypothesis: FMXIN002 will terminate anaphylactic reactions as effectively-or more rapidly-than IM epinephrine, as measured by clinical parameters.

DETAILED DESCRIPTION:
Study Procedures

1. Informed Consent: Participants will sign consent forms.
2. Food Challenge: Subjects will undergo routine diagnostic oral food challenges (OFC) relevant to their suspected allergens.
3. Assessment: At the first signs of allergic symptoms, a physician will assess the subject.
4. Treatment Criteria: If a Grade II or III anaphylactic reaction occurs, the participant will receive either:

   A). Intranasal spray of epinephrine FMXIN002 4mg + placebo saline injection B). Intranasal spray of placebo + intramuscular epinephrine injection (Adrenalin 0.5mg)

   One administration will always be epinephrine; the other, placebo.
5. Randomization: 1:1 between the 2 study arms.
6. Exclusion from Trial Treatment: Severe reactions or physician discretion may warrant standard care (IM epinephrine 0.5 mg) without study drug.
7. Blinding: Double-blinded setup with pre-prepared, numbered envelopes containing randomized treatment kits (nasal spray + injection).
8. Supportive Treatment: All participants will receive antihistamines (Fenistil drops + fexofenadine 180 mg or desloratadine 5 mg). Inhaled bronchodilators (e.g., Ventolin) will be provided for respiratory symptoms as needed.
9. Monitoring: Assessments at baseline, symptom onset, and at 3, 5, 10, 15, 30, and 90 minutes post-treatment. Vital signs and system-based symptom assessments will be recorded (Appendix 3).
10. Rescue Therapy: If no improvement in 3-5 minutes, a second IM epinephrine dose (0.5 mg) will be given. Further treatment will follow standard anaphylaxis protocols
11. Discharge: Participants with symptom resolution by 90 minutes will be discharged.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years, any gender
* Documented or suspected food allergy (based on IgE level or clinical history)
* Development of Grade II or III reaction during OFC

Exclusion Criteria:

* Age <18 or >40
* Poorly controlled asthma (FEV1 < 80% or frequent symptoms)
* Active eosinophilic esophagitis
* Pregnancy or risk of pregnancy
* Mild (Grade I) or very severe (Grade IV) reactions during OFC
* Decline to participate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-07-12 (Estimated)

PRIMARY OUTCOMES:
Skin system anaphylaxis symptoms | 0-90 minutes after drug administration
  Severity grading system for acute allergic reactions. Skin system, severity score 0 (=no reaction) to 5(= severe reaction), based on the Delphi study, 2021
Mucosal system anaphylaxis symptoms | 0-90 minutes after drug administration
  Severity grading system for acute allergic reactions, mucosal system, severity score 0 (=no reaction) to 5(= severe reaction), based on the Delphi study, 2021
Gastrointestinal system anaphylaxis symptoms | 0-90 minutes after drug administration
  Severity grading system for acute allergic reactions, gastrointestinal system, severity score 0 (=no reaction) to 5(= severe reaction), based on the Delphi study, 2021.
Respiratory system anaphylaxis symptoms | 0-90 minutes after drug administration
  Severity grading system for acute allergic reactions, respiratory system, severity score 0 (=no reaction) to 5(= severe reaction), based on the Delphi study, 2021.
Total anaphylaxis severity score | 0-90 minutes after drug administration
  Severity grading system for acute allergic reactions, Combined systems, anaphylaxis score 0 (=no reaction) to 5(= severe reaction), based on the Delphi study, 2021.
Vital signs: Blood pressure | 0-90 minutes after drug administration
  Systolic and diastolic blood pressure by a blood pressure cuff
Vital signs: pulse rate | 0-90 minutes after drug administration
  heart rate by pulse rate measurement
Vital signs: oxygen saturation | 0-90 minutes after drug administration
  % oxygen saturation measurement using oxygen monitor

SECONDARY OUTCOMES:
Need for a second epinephrine dose | 0-90 minutes after drug administration
  Number of patients needed a second dose, by Adrenalin IM injection
Adverse events | 0-90 minutes after drug administration
  Any treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Elizur, Prof., Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Shamir Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No